CLINICAL TRIAL: NCT00743938
Title: A Double-Blind, Randomized, Parallel Two-Arm Phase II Trial of BMS-690514 Versus Erlotinib in Previously Treated NSCLC Patients
Brief Title: A Comparison Between BMS-690514 and Erlotinib in Patients Who Were Previously Treated for NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA187-017; EUDRACT #: 2008-004691-44
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — BMS-690514; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: BMS-690514
- B2 (Active Comparator)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: BMS-690514 — Tablets, Oral, 200 mg, once daily, Until disease progression or toxicity
  Other Names: panHER
  Arms: A1
Drug: Erlotinib — Capsules, Oral, 150 mg, once daily, Until disease progression or toxicity
  Other Names: Tarceva
  Arms: B2

SUMMARY:
The purpose of this study is to improve disease control and survival for patients who were treated with chemotherapy using BMS-690514 over erlotinib

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS of 0 or 1
* Histologically confirmed NSCLC
* Adequate amount of tumor (archived or fresh) for biomarker evaluation
* Received one to two regimens of chemotherapy (with at least one platinum-containing)
* Serum creatinine of less than 1.0 mg/dL or a 24 hour creatinine clearance of greater than 60 mL/min
* Stable control of blood pressure on agents other than calcium channel blockers
* Women of child-bearing potential must avoid pregnancy or maintain adequate contraception
* Must be able to swallow pills and take the medications at the same time every day on an empty stomach

Exclusion Criteria:

* ECOG PS 2 or greater
* Women unwilling to avoid pregnancy or use adequate contraception
* Symptomatic brain metastases
* Recent history of TIA, CVA, or thrombotic/thromboembolic event (within 6 months)
* History of hemoptysis greater than 10 mL/day
* Significant cardiovascular disease
* Uncontrolled diarrhea, Crohn's disease, ulcerative colitis, or any malabsorptive disease
* History of use of other TKIs
* Uncontrolled hypertension
* HIV+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To compare the progression-free survival of patients on BMS-690514 with those on erlotinib | CT/MRI at baseline and every 6 weeks for 36 weeks

SECONDARY OUTCOMES:
To compare the overall survival between BMS-690514 and erlotinib | 15 months
To estimate the overall response rate of BMS-690514 or erlotinib | 15 months
To estimate the tumor size change and PFS rate at 6 weeks | 6 weeks
To assess safety and tolerability of BMS-690514 and erlotinib | 15 months
To estimate the association between efficacy and EGFR copy as measured by FISH for both BMS-690514 and erlotinib | 15 months
To obtain samples for population pharmacokinetics for BMS-690514 in previously treated NSCLC patients | Days 1,8,15, 29

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (28):
- United States (9):
  - Yale University School Of Medicine, New Haven, Connecticut
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Mass General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Piedmont Hematology Oncology Associates, Pllc, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Hema/Oncology Assoc. Of Nepa, Dunmore, Pennsylvania
  - Cancer Center Of The Carolinas, Greenville, South Carolina
- Argentina (5):
  - Local Institution, Bahía Blanca, Buenos Aires
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, La Rioja, La Rioja Province
- Canada (2):
  - Local Institution, Montreal, Quebec
  - Local Institution, Sherbrooke, Quebec
- France (5):
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Local Institution, Otwock, Poland
- South Korea (2):
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Vizcaya
- Local Institution, Taipei, Taiwan

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx